CLINICAL TRIAL: NCT06953219
Title: Investigation of the Relationship Between 2D:4D Ratio and Proprioception
Brief Title: Relationship Between 2D:4D Finger Ratio and Proprioception
Status: Completed | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Onur Engin, Dr., Izmir Democracy University
Other Study IDs: 2025/405
Record Dates: First submitted 2025-04-22; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Proprioception
Keywords: digit ratio; proprioception

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- assessment group: Finger length measurements(second digits and fourth digit) were made with acaliper. Range of motion (ROM) and joint position error measuremenst were made with a CROM device. Joint position error is assessed with neutral head positioning test and target head positioning test.

SUMMARY:
Background: 2D:4D ratio (the ratio of the length of the second digit to the length of the fourth digit) has been reported to be associated with muscle strength and physical performance, numerical competencies, spatial skills and cognitive abilities. However, the relationship between 2D:4D ratio and proprioception is not well-known, which was therefore aimed at investigating in current study. Methods: 2D:4D ratio (electronic digital calliper) and proprioception (Join position error is measure with Cervical Range of Motion instrument) were assessed in all individuals (n=35.7 ± 11.2 years).

DETAILED DESCRIPTION:
2nd (index) and 4th (ring) finger ratio, index finger (2nd finger) length to ring divided by the length of the fourth finger (4th finger) and is referred to in the literature as the "2D:4D ratio". The reference points for 2D:4D ratio measurement are the midpoint of the proximal ventral flexion bend of the finger and the distal end of the finger. 2D:4D ratio is a function of prenatal exposure to testosterone and estrogen levels and shows gender-related differences. A low 2D:4D ratio indicates that prenatal testosterone levels are high and estrogen levels are lower, while a high 2D:4D ratio indicates lower testosterone and higher estrogen exposure. For example, men's index fingers (2D) are longer than their ring fingers (4D), while in women the second finger is usually significantly shorter than or slightly shorter than or equal to the fourth finger. In recent years, several studies have been conducted on the biological and behavioral associations with the 2D:4D ratio. For example, a low 2D:4D ratio is often associated with increased physical strength, athletic performance, and risk-taking behavior, while a high 2D:4D ratio is associated with traits such as empathy and language skills. Proprioception, which refers to the ability to sense joint and body movement, as well as the movement of the body or body segments, is defined as the perception of its position in space. Proprioception plays a critical role for balance, coordination, and motor control. The 2D:4D ratio, influenced by hormonal changes, may affect proprioceptive functions, such as motor skills and hand-eye coordination. Some studies have found that individuals with low 2D:4D ratios perform better on tasks involving mental rotation of two- and three-dimensional objects. Testosterone exposure during the prenatal period is thought to increase the development of the right hemisphere of the brain. Proprioception, a person's ability to perceive body position and movements, can also be significantly influenced by the 2D:4D ratio. The ratio is influenced by both genetic factors and prenatal environmental influences. For example, human tool manipulation in the course of evolution contributed to the differentiation and specialization of brain areas associated with sensory and motor skills. Some research suggests that a low 2D:4D ratio may be linked to stronger motor skills and a better proprioceptive sense. This is because prenatal testosterone levels affect motor control and nervous system development, influencing hand-eye coordination. For example, individuals with a low 2D:4D ratio may show improved hand-eye coordination and performance in tasks requiring fine motor control. A study examined the relationship between hand morphometry (including 2D:4D ratio) and proprioception and found that haptic perception was closely related to proprioception. Lower 2D:4D ratios were associated with better physical strength and precise motor control. Additionally, lower 2D:4D ratios have shown an association with better arithmetic, visual, and spatial skills. However, there are no available studies that directly address the relationship between proprioception and the 2D:4D ratio. Therefore, more research is needed to understand the connection between proprioception and 2D:4D ratio. The aim of this study is to investigate the relationship between the 2D:4D ratio and proprioception in adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Agreeing to participate in the study.

Exclusion Criteria:

* Individuals who have scars, finger deformities, and/or surgical interventions that would prevent accurate measurement of the 2D:4D ratio
* Congenital hand anomalies
* History of trauma involving the hand or cervical region were excluded from the study.
* Having sensory loss or severe neurological disorder that would affect proprioception

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult individuals aged between 18 and 65 years, who volunteered to participate in the study. Participants had no sensory loss or severe neurological disorders affecting proprioception. Individuals with hand or cervical trauma history, congenital hand anomalies, or any condition preventing accurate 2D:4D measurement were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-03-24 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Finger length measurement and 2D:4D ratio calculation | baseline
  The lengths of the second (2D) and fourth (4D) fingers on each hand were measured using an electronic digital caliper with a precision of 0.01 millimeters. Measurements were taken on the palmar surface of the hand, extending from the distal tip of the finger to the basal crease at the proximal end of the digit.The 2D:4D ratio was calculated separately for the right and left hands. To enhance the accuracy of the 2D:4D ratio measurements, each finger was measured three times during a single assessment session by the same investigator. The repeated measurements were not taken consecutively; instead, at least one other hand was measured between the first and second measurements of any given hand. This procedure was implemented to minimize the potential influence of recall bias on subsequent measurements.
Cervical Range of Motion | baseline
  The cervical range of motion measurement was performed using a Cervical Range of Motion (CROM) device, which is a reliable and valid tool. The CROM unit is a mechanical instrument that measures cervical ranges by combining a magnetic reference with standard inclinometers. The individuals were told to sit comfortably with their hands on the armrest and their backs straight on the chair. The CROM unit was secured on the individuals' head by the physiotherapist. The CROM unit's magnetic yoke is positioned squarely around the neck with its arrow pointing directly north. Afterwards, physiotherapist asked individuals to perform cervical range of motion in all three directions: flexion- extension, lateral flexion and rotation.The maximum range of cervical flexion, extension, left and right rotation, and left and right lateral flexion was measured three times and averaged.
Repositioning to neutral head position (NHP) | baseline
  For the NHP assessment, the individuals were asked to keep their head in the neutral head position, with their eyes closed. The deviations from the neutral (0) position in the sagittal (flexion-extension), frontal (lateral flexion), and transverse (rotation) planes were recorded using the CROM device.
Repositioning the head to a predetermined reference point (Target Head Position, THP) | baseline
  For the assessment of THP, the target position will be defined as half of the maximum active range of motion measured during a standard cervical joint mobility assessment. While the patient's eyes are covered with an eye mask, the head will first be slowly positioned by the physiotherapist to the predetermined target angle and held in this position for five seconds for the patient to perceive. Subsequently, the head will be moved away from the target position, and the patient will be asked to actively reposition it to the original target. Each measurement will be repeated three times, and the mean deviation from the target angle will be recorded. Measurements will be conducted separately for flexion, extension, right rotation, left rotation, right lateral flexion, and left lateral flexion

CONTACTS AND LOCATIONS:
Overall Officials: Onur Engin, Assist Prof, Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Izmır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It was deemed appropriate to keep the data of the individuals participating in the study confidential